CLINICAL TRIAL: NCT00925197
Title: Patient INR Self-Testing Program Improves the Quality of Oral Anticoagulant Therapy After Mechanical Heart Valve Replacement
Brief Title: Patient International Normalised Ratio (INR) Self-Testing Program
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Abbott Medical Devices (Industry); Roche Diagnostics GmbH (Industry); HemoSense (Industry)
Responsible Party: Patrick Lacarin, CHU Clermont-Ferrand
Allocation: Randomized | Masking: None
Other Study IDs: CHU-0054
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Mechanical Aortic and/or Mitral Valve Replacement Operation
Keywords: anticoagulation; fluindione; patient self-testing; coaguchek; inratio; Post operative antivitamin K therapy

INTERVENTIONS:
Other: INR self-testing program

SUMMARY:
The aims of the study are to prove correlation between laboratory and patient self-testing (PST) measurements, estimation of INR variability within a target therapeutic zone and frequency of hemorrhagic and/or thromboembolic events after mechanical heart valve replacement.

DETAILED DESCRIPTION:
This is the first French, prospective, randomised, single centre study, comparing patient self-testing (PST) of international normalised ratio (INR), with conventional laboratory monitoring. Aims of the study are to prove correlation between laboratory and PST measurements, estimation of INR variability within a target therapeutic zone and frequency of hemorrhagic and/or thromboembolic events after mechanical heart valve replacement.

Patients (206) were postoperatively, randomly, consecutively included (2004 - 2008): 103 patients in each group, with a one year follow-up. Two INR control devices were selected: Coaguchek® (Roche) and INRATIO® (Hemosense).

ELIGIBILITY:
Inclusion Criteria:

* adults
* patients fitted with one or more mechanical heart valves either alone or in combination with myocardial revascularization
* oral anticoagulant treatment
* patients with social security cover
* written informed consent signed by both patient and investigator
* able to be followed up during 12 months

Exclusion Criteria:

* refusal of participation in the study
* Participation in another clinical study
* Patient is pregnant or nursing
* Life expectancy less than three months
* Contra-indication of to an A.V.K treatment
* Difficult comprehension of the French language
* Patients unable to master the self-monitoring procedures
* Individuals under judicial control or enquiry
* Patients on dialysis Patients with incomplete understanding of instructions
* Blind patients and those unable to read

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2004-05; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Hemorrhagic events and thromboembolic events | after mechanical heart valve replacement

SECONDARY OUTCOMES:
Correlation of laboratory INR and device INR control | after mechanical heart valve replacement

CONTACTS AND LOCATIONS:
Overall Officials: Kasra Azarnoush, MD, Principal Investigator — University Hospital, Clermont-Ferrand

REFERENCES:
- [Derived] Azarnoush K, Dorigo E, Pereira B, Dauphin C, Geoffroy E, Dauphin N, D'Ostrevy N, Legault B, Camilleri L. Mid-term results of self-testing of the international normalized ratio in adults with a mechanical heart valve. Thromb Res. 2014 Feb;133(2):149-53. doi: 10.1016/j.thromres.2013.09.013. Epub 2013 Sep 16. PMID 24112749